CLINICAL TRIAL: NCT05210231
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Rotator Cuff Fatigue. A Randomized, Sham-controlled, Double-blind, Crossover Study.
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Rotator Cuff Fatigue.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gran Rosario (Other)
Responsible Party: Principal Investigator, Mauro Barone, Principal Investigator, University of Gran Rosario
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: tDCS and Rotator Cuff
Record Dates: First submitted 2022-01-25; First posted 2022-01-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-03

CONDITIONS: Asymptomatic Condition
Keywords: Brain stimulation; tDCS; Fatigue; Rotator cuff
MeSH Terms: conditions — Asymptomatic Diseases; Fatigue | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active anodal tDCS (Experimental): The direct electric current will be applied through a pair of sponges humidified with saline solution (150 mMols of NaCl diluted in water Milli-Q) on the electrodes (35 cm2). The electrodes (anode and cathode) will be connected to a continuous electric stimulator (Model: Microestim Foco Research, Brand: NKL, Souza Cruz, Brusque - SC, Brazil), with one energy battery (9 V) and will be mounted in accordance with the International 10-20 EEG System. For anodal polarity stimulation over the left TC, the anodal electrode will be placed over the scalp on the T3 area located at 40% of the distance on the left from the Cz point. The cathode electrode will be placed over the contralateral supraorbital area (Fp2). Thereafter, a constant electric current of 2 mA will be applied for 20 min.
  Interventions: Other: Transcranial Direct Current Stimulation
- Sham anodal tDCS (Sham Comparator): The direct electric current will apply through a pair of sponges humidified with saline solution (150 mMols of NaCl diluted in water Milli-Q) on the electrodes (35 cm2). The electrodes (anode and cathode) will be connected to a continuous electric stimulator (Model: Microestim Foco Research, Brand: NKL, Souza Cruz, Brusque - SC, Brazil), with one energy battery (9 V) and will be mounted in accordance with the International 10-20 EEG System. For the sham condition, the electrodes will be placed at the same positions as for the anodal tDCS. However, the stimulator will turn off after 30 s of stimulation. As a result, subjects will report the same sensory feelings from the beginning of the real tDCS conditions, specifically itching and tingling feelings on the scalp for the first few seconds of tDCS, but not thereafter, whether or not the stimulation will continue or stop.
  Interventions: Other: Transcranial Direct Current Stimulation

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation — The direct electric current will be applied through a pair of sponges humidified with saline solution (150 mMols of NaCl diluted in water Milli-Q) on the electrodes (35 cm2). The electrodes (anode and cathode) will be connected to a continuous electric stimulator (Model: Microestim Foco Research, Brand: NKL, Souza Cruz, Brusque - SC, Brazil), with one energy battery (9 V) and will be mounted in accordance with the International 10-20 EEG System. For anodal polarity stimulation over the left TC, the anodal electrode will be placed over the scalp on the T3 area located at 40% of the distance on the left from the Cz point. The cathode electrode will be placed over the contralateral supraorbital area (Fp2). Thereafter, a constant electric current of 2 mA will be applied for 20 min.

SUMMARY:
The aim of this study will be to determine the effects of active tDCS on rotator cuff fatigue. This study will be a randomized, double-blind, sham-controlled, cross-over clinical trial based on non-probabilistic sampling for convenience, comprising a sample of 20 active asymptomatic subjects of all genders and aged between 18 and 35 years old. Subjects will be recruited via social networks, WhatsApp and emails and must be currently engaged in moderate physical activity (assessed by the IPAQ questionnaire) and asymptomatic at the time of assessment. In addition, participants will be asked not to perform any type of strenuous exercise and do not drink alcoholic or caffeinated beverages during the time the work is performed. The study will consist of three sessions, with an interval of 72 hours between them.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 18 to 35 years, all genders.
* Healthy subjects
* Moderate physical activity (evaluated by IPAQ questionnaire)
* Do not perform any exhausting exercise and do not drink alcoholic or caffeinated beverages during the time the work is performed.

Exclusion Criteria:

* Subjects with trauma in the last three weeks or previous surgeries on the upper extremity, patients with pre-existing neurological or rheumatic conditions, pregnancy, medical history of epilepsy the convulsive event, subjects under analgesic drug treatment or have ingested drugs with central action in the last 72 hours.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Time to Exhaustion (TTE) | At baseline, after 3 and 6 days
  To assess endurance performance, participants will perform a submaximal isometric time to exhaustion (TTE) task of the shoulder external rotator muscles at 50% of their maximal voluntary contraction (MVC), which will be performed during each visit. During the TTE each participant will receive visual feedback on a computer monitor showing the target force. The task will finish when their force is below the required target value for more than 3 s. None of the participants will be aware of the time elapsed during the test and results of all the sessions will be provided only after the completion of all visits. Participants' perception of effort will be measured using the RPE scale (Borg, 1998) every 20 s of the TTE task. Leg muscle pain will be assessed every 20 s by using the Numerical Pain Rating Scale (NPRS).
Change in Maximum Voluntary Contraction (MVC) | At baseline, after 3 and 6 days
  After a brief standardized warm-up with submaximal isometric contractions, all participants will perform a 6 seconds MVC of infraspinatus muscle. For the MVC, subjects will be standing, with the shoulder in adduction position and the elbow flexed at 90°. The record will be evaluated by a load cell S200 (Miotec™, Porto Alegre, Brazil). The MVC produced during this test will be used to calculate the participants' 50% MVC used in the subsequent TTE task of that visit.
Change in Rating of Perceived Exertion (RPE) | At baseline, after 3 and 6 days
  Borg rating of perceived exertion (RPE) is an outcome measure scale used in knowing exercise intensity prescription. The RPE will be evaluated using the BORG CR10 scale, its ranges are from "0" (no exertion) to "10" (maximum effort). The RPE will be evaluated using the BORG CR10 scale, its ranges are from "0" (no effort) to "10" (maximum effort). The perception of the effort of the participants will be measured every 20 s during the TTE task.

SECONDARY OUTCOMES:
Change in Global Rating of Change Scale (GRCS) | After 3 and 6 days
  For the Global Rating of Change Scale, in the second and third visit, subjects will be asked about their perception of change in relation to the endurance task relative to their status at the first visit.
Change in Electromyographic recordings (sEMG) | At baseline, after 3 and 6 days
  Surface electromyography (sEMG) assessment will be performed on the infraspinatus and deltoid muscles, using an acquisition module with four analog channels (Miotec™, Biomedical Equipments, Porto Alegre, Brazil). The conversion from analog to digital signals will be performed by an A/D board with 16-bit resolution input range, sampling frequency of 2 kHz, common rejection module greater than 100 dB, signal-noise ratio less than 03 μV Root Mean Square and impedance of 109 Ω. The sEMG signals will be recorded through surface Ag/AgCl electrodes (Meditrace™, Canada) with a centre-to-centre distance of 2 centimeters, in a parallel orientation to the underlying muscle fibers. A ground electrode will be placed in the lateral epicondyle of the contralateral arm The skin will be shaved and cleaned using alcohol swabs, following standardized guidelines. A fatigue study will be carried out using a frequency analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Mendoza, MsC, Principal Investigator — University of Gran Rosario
Locations (1):
- University of Gran Rosario, Rosario, Santa Fe Province, Argentina